CLINICAL TRIAL: NCT00477477
Title: Nutritional Treatment of Overweight Adolescents With Cardiovascular Risk Factors
Brief Title: Nutritional Treatment of Overweight Adolescents With Cardiovascular Risk Factors (PowerUp)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment and lack of funds.
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sarah D. de Ferranti, Assistant Professor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-01-0020; K23HL085308 (NIH)
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Childhood Obesity; Dyslipidemia; Insulin Resistance; Hypertension
Keywords: overweight; metabolic syndrome; adolescent; cardiovascular; risk factors; hypertension; dyslipidemia; inflammation; coagulopathy
MeSH Terms: conditions — Pediatric Obesity; Dyslipidemias; Insulin Resistance; Hypertension; Overweight; Metabolic Syndrome; Inflammation; Hemostatic Disorders | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Low glycemic load diet
  Interventions: Other: Diet
- 2 (Active Comparator): Low fat diet
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Low glycemic load diet prepared/delivered for 8 weeks, and counseled for 4 more months. Daily multivitamin.
  Arms: 1
Other: Diet — Low saturated fat diet prepared/delivered for 8 weeks, and counseled for 4 more months. Daily multivitamin.
  Arms: 2

SUMMARY:
This study is designed to evaluate the efficacy of two diets, a low glycemic load diet and a low saturated fat diet, in the treatment of adolescents with some heart disease risk factors associated with being overweight, such as high blood pressure, pre-diabetes, and cholesterol problems. The objective of the study is to determine which diet improves these risk factors more. The design of the study is a modified feeding study, which requests that the participants eat all and only the food provided by the study for 8 weeks, most days per week. Dietary counseling by phone will continue between 2 and 6 months of the study and the effects of this maintenance period will be assessed at 6 months time.

DETAILED DESCRIPTION:
The prevalence of obesity and overweight among children is high, and increasing. Metabolic syndrome, a recently recognized consequence of obesity, is known to confer an elevated risk for cardiovascular (CV) disease and diabetes type 2 in adults. The primary treatment for metabolic syndrome is lifestyle modification, including dietary changes. However, little is known about how dietary composition, as distinct from decreased caloric intake and weight loss, alters metabolic syndrome abnormalities in children. Moreover, the optimal pediatric nutritional strategy for prevention and treatment of metabolic syndrome is unknown. The overall goal of this research protocol is to evaluate two nutritional approaches to pediatric metabolic syndrome in post-pubertal overweight adolescents, a low saturated fat diet and a low glycemic load (GL) diet. The design of the protocol is a short-term, modified feeding study that evaluates the efficacy of these two nutritional approaches with equal weight loss goals. Outcome measures will include the percent changes from baseline to the end of the intervention period (8 weeks) in metabolic abnormalities, inflammatory cytokines and adipokines, and non-invasive tests of vascular function. Metabolomic profiles are measured at baseline and 8 weeks in a subset of the participants.

To facilitate compliance and adherence, participants chose from a menu of food choices and food will be delivered to participants homes to supply most of the meals and snacks participants consume. Participants will receive weekly personal nutritional counseling to enhance compliance with frequent phone follow-up. Subsequent to the feeding portion of the intervention, participants are counselled by phone at least on a monthly basis and the effects of this maintenance phase is measured at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8 to 17 years old
* Overweight, defined as BMI ≥ 85th%tile for age and gender
* At least two CV risk factor typical of the metabolic syndrome including insulin resistance, high or borderline blood pressure, low HDL, high TG
* Insulin > 10 u/L
* Able to attend study visits once a week at participant's home, and eat meals provided by the Children's Hospital CTSA Boston MA as supplied for most meals and snacks
* Non-smoker
* Able to understand/speak English
* Informed consent to participate from a parent or legal guardian. Adolescents must also provide written assent to participate in the study.

Exclusion Criteria:

* Pre-existing physician diagnosis of a major medical illness or history of a major medical illness including but not limited to heart, kidney or liver disease, cancer, endocrinopathy including thyroid disorder, genetic syndrome or psychiatric illness, also including vasculitides such as Kawasaki disease or rheumatologic disorder; diabetes type I or II, evidence of severe fatty liver, hypertension requiring pharmacologic treatment, history of or current diagnosis of an major eating disorder
* Current or anticipated pregnancy
* Weight more than 275 lbs (125 kg)
* Abnormalities on initial screening assessment requiring pharmacotherapy urgent treatment, such as familial hyperlipidemia, end organ effects of hypertension, or metabolic abnormalities such as diabetes
* Taking any prescription medication or non-prescription substance that affects cholesterol levels, blood pressure, or insulin sensitivity (including but not limited to oral glucocorticoids, oral contraceptives, neuropsychiatric agents, anti-epileptics, HMG-CoA reductase inhibitors, bile acid binding cholesterol transport inhibitors among others) and the use of alcohol or illicit substances.
* Anticipated difficulty with participatory requirements of the study including food allergies, significantly restricted food preferences, or other difficulties as assessed by research staff.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2007-05; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | 8 weeks, 6 months

SECONDARY OUTCOMES:
Inflammation | 8 weeks, 6 months
dyslipidemia | 8 weeks, 6 months
blood pressure | 8 weeks, 6 months
coagulopathy | 8 weeks, 6 months
vascular function | 8 weeks, 6 months
liver function testing | 8 weeks, 6 months
Metabolomic profile | baseline, 8 weeks
  The metabolomic profile of a subset of the participants will be measured at baseline and 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah D. de Ferranti, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States